CLINICAL TRIAL: NCT03961451
Title: Number of Weekly Steps, Fatigue, Quality of Life, Well-being During Cancer Treatment: Impact of Recommendations Strengthened by the Provision of Web Interface and Tele-coaching.
Acronym: PODOMETRE
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: PODOMETRE-IPC 2015-028
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cancer, Treatment-Related
Keywords: pedometer
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group With Recommendations (GAR): Patients in the GAR group will receive several recommendations and will have access to an online tool to increase motivation to engage in physical activity.
  Interventions: Device: Podometer
- Control Group (GC): No recommendation given
  Interventions: Device: Podometer

INTERVENTIONS:
Device: Podometer — Patients will be equipped with pedometers for 8 weeks, all day and must complete the number of steps each day. They will have to complete online evaluation questionnaires regularly. The main objective is to correlate the level of physical activity with the level of fatigue, quality of life and well-being weekly during an anticancer treatment.

SUMMARY:
study to correlate this level of objective physical activity with the levels of fatigue and quality of life in cancer patient being treated.

DETAILED DESCRIPTION:
Study to objectify the level of physical activity of patients by a tool, often used in the global population: the pedometer. Several measurements per questionnaire also will be carried out repeatedly (weekly) in order to correlate this level of objective physical activity with the levels of fatigue and quality of life. The hypothesis we formulate is as follows: the number of weekly steps is negatively correlated with the level of fatigue, positively with the quality of life and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated, Medical Day Hospital / HAD

Exclusion Criteria:

* Inability to walk declared by an site medical doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cancer pathologies, all treatments. Provided that the patient is fit for walking.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Life satisfaction | 2 months
  Satisfaction With Life Scale (Blais et al, 1989, french-canadian validation, Revue Canadienne des Sciences du Comportement, 21(2), 210-223.)
Positive and negative affects measurement | 2 months
  Positive and Negative Affect Schedule (PANAS scales) (Caci et Baylé, 2007 First traduction in French, Congrès de l'Encéphale, Paris, 25-27 january 2007)
Fatigue | 2 months
  Multidimensional Inventory Fatigue : Gentile et al, 2003, Validation of the French multidimensional fatigue inventory (MFI 20), Eur J Cancer Care)
Quality of Life | 2 months
  European Organisation for Research and Treatment of Cancer Questionnaire Quality of Life version 30

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cappiello, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Villaron C, Cury F, Eisinger F, Cappiello MA, Marqueste T. Telehealth applied to physical activity during cancer treatment: a feasibility, acceptability, and randomized pilot study. Support Care Cancer. 2018 Oct;26(10):3413-3421. doi: 10.1007/s00520-018-4191-4. Epub 2018 Apr 19. PMID 29675546